CLINICAL TRIAL: NCT06517290
Title: Evaluation of the Risk of Infection During Fever in Labor
Acronym: FEVERY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240875
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Fever; Labor
Keywords: Fever; Labor; Puerpueral infection; Anti-Bacterial Agents
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fever during labor
  Interventions: Other: Non applicable
- Child
  Interventions: Other: Non applicable

INTERVENTIONS:
Other: Non applicable — Non applicable

SUMMARY:
* Fever during labor affects more than 8% of parturients. It is a heterogeneous entity and can be due to an infectious process, a side effect of a drug, or to labor itself (physiological hyperthermia).
* It has been the subject of several retrospective studies and a few prospective studies with varying methodologies, definitions, and inclusion criteria. None have proposed a combined obstetric, neonatal, infectious disease, and microbiological analysis.
* It raises concerns about the possibility of an emerging maternal (obstetric or otherwise) and/or fetal infection.
* Analysis of the available literature does not clarify the exact frequency of these infections or the predictive factors for their occurrence.
* It often justifies systemic antibiotic therapy, the modalities and benefits of which have never been evaluated.

The investigators aim to conduct a prospective multicenter study to analyze fever during labor with a combined obstetric, infectious disease, pediatric, and microbiological perspective.

DETAILED DESCRIPTION:
The primary objective of this study is to analyze the causes of fever during labor by categorizing them into 3 etiological categories:

1. Fever indicative of maternofetal infection: potentially early intrauterine infection leading to proven or probable early-onset neonatal bacterial infection, endometritis, or maternal sepsis.
2. Fever indicative of maternal infectious pathology outside the obstetrical field (e.g., pyelonephritis, influenza, COVID, etc.).
3. Fever of non-infectious origin.

Secondary objectives include:

* Describing the epidemiology and local ecology of bacterial infections.
* Identifying predictive factors for each category (obstetrical infection, non-obstetrical infection, and non-infectious fever) when fever occurs during labor.
* Evaluating the maternal and neonatal prognosis of mother-child pairs who do not receive antibiotic treatment according to local protocols (e.g., in cases of fever below a threshold value).

Depending on the results and sample size, the study will also attempt to evaluate the maternal and neonatal prognosis of mother-child pairs in cases where fever is attributed to maternofetal infectious causes (category 1) according to the antibiotic management strategy for fever during labor at each center.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least more than 37 weeks
* Who have not opposed the collection of their health data for the purposes of studies and analyzes
* In work between 07/01/2023 and 06/01/2024
* Admitted to the work room at Port Royal, Necker Sick Children or Trousseau
* With fever defined as a tympanic temperature > 38°C at least 2 times at 10 min intervals during labor.

Exclusion Criteria:

* Pregnant women :
* < 37NT
* express their opposition to the collection of their data for research purposes
* minors or under legal protection
* context of medical termination of pregnancy or fetal death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women admitted to any of the three public university hospitals in Paris namely Port Royal, Necker - enfants maladies, Trousseau (AP-HP).
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Percentage of maternal-fetal infections | Up to 6 months
  intrauterine infection possibly responsible for early neonatal bacterial infection (proven or probable), endometritis, maternal sepsis
Percentage of proven maternal bacterial infections | Up to 6 months
  (non-obstetric, intrauterine, endometritis)
Percentage of proven and probable early neonatal infections | Up to 6 months

SECONDARY OUTCOMES:
occurrence of proven or probable early neonatal infection | Up to 6 months
  Maternal and neonatal prognosis
occurrence of endometritis | Up to 6 months
  Maternal and neonatal prognosis
Occurrence of maternal sepsis | Up to 6 months
  Maternal and neonatal prognosis
Occurrence of serious accident III or IV linked to the prescription of antibiotics | Up to 6 months
  Maternal and neonatal prognosis
Percentage of antibiotic therapy | Up to 6 months
  Type of care by category

CONTACTS AND LOCATIONS:
Overall Officials: Caroline CHARLIER, MD, PhD, Principal Investigator — Infectious diseases department of Cochin hospital
Locations (3):
- France (3):
  - APHP - Trousseau Hospital - Gynecology-Obstetrics-Maternity, Paris, IDF
  - AP-HP - Cochin Hospital - Maternity, Paris, IDF
  - APHP - Necker Hospital - Maternity, Paris, IDF

IPD SHARING:
Plan to Share IPD: No